CLINICAL TRIAL: NCT06115031
Title: Effect of Remimazolam Versus Propofol Anesthesia on Postoperative Delirium in Neurosurgical Patients: A Randomised, Controlled, Noninferiority Trial
Brief Title: Remimazolam vs. Propofol: Impact on Postoperative Delirium in Neurosurgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jiseon Jeong, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMC 2023-08-135
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; Remimazolam; Total intravenous anesthesia; Neurosurgery
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): General anesthesia using continuous infusion of intravenous remimazolam and remifentanil. Remimazolam will be used for maintenance of general anesthesia and adjusted between 0.6-2mg/kg/hr until the end of surgery.
  Interventions: Drug: Remimazolam
- Propofol (Active Comparator): General anesthesia using target-controlled infusion of intravenous propofol and remifentanil. Propofol will be adjusted maintaining the BIS between 40-60 until the end of surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — General anesthesia will be induced and maintained using continuous infusion of intravenous remimazolam.
  Other Names: byfavo inj
  Arms: Remimazolam
Drug: Propofol — General anesthesia will be induced and maintained using target-controlled infusion of intravenous propofol.
  Other Names: Fresofol
  Arms: Propofol

SUMMARY:
The investigator aimed to evaluate the incidence of postoperative delirium after remimazolam-based total intravenous anestheisa (TIVA) compared to the propofol-based TIVA in patients undergoing neurosurgery.

DETAILED DESCRIPTION:
Remimazolam, a short-acting benzodiazepine, has recently gained approval for use in the induction and maintanance of general anesthesia. In American Society of Anesthesiologists (ASA) physical status class I and II patients undergoing general anesthesia, the remimazolam-based TIVA has shown comparable efficacy to propofol-based TIVA while demonstrating a superior safety profile. Remimazolam has exhibited a lower incidence of hypotension, reduced vasopressor requirements, and fewer instances of bradycardia compared to the propofol-based TIVA.

The use of benzodiazepine has been associated with an increased risk of postoperative delirium, but there is currently no randomized controlled trial investigating the relationship between remimazolam, a new short-acting benzodiazepine, and postoperative delirium. Therefore, the investigators designed this prospective, randomized, double-blinded, active comparator-controlled, non-inferiority trial to investigate the incidence of postoperative delirium after remimazolam-based TIVA compared with propofol-based TIVA in neurosurgery patients.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesia (ASA) class I - III

Exclusion Criteria:

* Severe respiratory, cardiovascular, or hepatic disease (child-pugh C)
* Dependency on psychiatric drugs or alcohol
* Severe sensory impairments that impede communication
* Preoprative delirium
* Hypersensitivity, allergies, or contraindication to the study drugs.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | assessed up to postoperative day 5 or patient discharge, whichever came first
  The occurence of postoperative delirium will be assessed twice a day using confusion assessment method for the intensive care unit (CAM-ICU) and 3-minute diagnostic assessment for CAM-defined delirium (3D-CAM).

SECONDARY OUTCOMES:
Onset of postoperative delirium | From the end of surgery until the date of first diagnosis of delirium or discharge, whichever came first, assessed up to postoperative day 5
  The time of initial diagnosis of postoperative delirium
Delirium subtypes | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  Hypoactive/hyperactive/mixed
Severity of postoperative delirium | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  Severity of postoperative delirium will be assessed twice a day using DRS-R-98 (delirium rating scale-revised-98)
Duration of postoperative delirium | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  Duration of postoperative delirium will be assessed twice a day
Subsyndromal delirium | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  Presence of any CAM features with absence of full syndromal delirium
Delirium symptoms | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  Subsyndromal delirium plus syndromal delirium
The proportion of valid delirium assessment | assessed twice a day up to postoperative day 5 or patient discharge, whichever came first
  The percentage of valid delirium assessments (per patient) that did not involve coma or stupor out of a total of 14 delirium assessments.
Intensive care unit (ICU) admission with endotracheal intubation after surgery | assessed up to postoperative day 5 or patient discharge, whichever came first
  Percentage of the patients who were not extubated in the OR and transferred to the ICU
Emergence agitation | within 30 min after extubation
  defined as Richmond Agitation-Sedation Scale ≥+1
Postoperative pain score | assessed once a day up to postoperative day 5 or patient discharge, whichever came first
  Pain level will be assessed using numeric rating score (NRS)
Opioid consumption | assessed once a day up to postoperative day 5 or patient discharge, whichever came first
  The amount of opioid consumption will be coverted to parenteral morphine equivalent dose (MED).
Intraoperative awareness | at postoperative day 0
  Intraoperative awareness will be assess using Modified brice questionnaire.
Undesirable patient movement | Intraoperative period
  Undesirable movement of patient during surgery
Potential adverse event | From the beginning of anesthesia until 24 hours after surgery
  hypotension, hypertension, bradycardia, tachycardia, desaturation, teeth injury, laryngeal spasm, allergic reaction, other arrhtymia, cardiac events, pruritis, nausea, vomiting etc
Perioperative serious adverse events | rom date of randomization until 24 hour after surgery
  Serious adverse events are adverse events that result in hospitalization or prolong hospitalization, cause persistent or significant disability, are life-threatening, or result in death.
Postoperative complication | Until 30 day after surgery
  assessed by Clavien-Dindo classification Data are presented as the proportion of patients with 1 or more events (edema, vasospasm, rebleeding, seizures, and/or ischemia, etc..)
Length of stay in ICU after surgery | from the day of surgery to the time of patient discharge from ICU, assessed up to 3 months after surgery
  days
Length of stay in hospital after surgery | from the day of surgery to the time of patient discharge, assessed up to 3 months after surgery
  days
Acute kidney injury (AKI) after surgery | within 1 week after surgery
  AKI assessed by KDIGO criteria
Myocardial injury after non-cardiac surgery (MINS) | within 1-month after surgery
  MINS assessed by high-sensitive TnT
Fall | 3-month after surgery
  the incidence of postoperative fall-down and associated injury (presence of fracture)
Postoperative cognitive dysfunction | 3-month after surgery
  assessed by T-MOCA (Montreal Cognitive Assessment) using telephone interview
Functional status | 3-month after surgery
  assessed using bartel activity of daily living (ADL) index
Death | during hospitalization (up to day 30), within 1 year after surgery (3, 6, and 12-month after surgery)
  All-cause mortality

OTHER OUTCOMES:
Postoperative nausea and vomiting (PONV) | within 3 days after surgery
  PONV substudy are pre-planned non-inferioirty substudy for this main trial. In addition to the data collected as part of the main trial, patients enrolled into the PONV substudy were assessed the frequency and severity of nausea and vomiting, and frequency of antiemetic administration using validated questinnaire.
Subgroup analysis of delirium incidence assessed by CAM-ICU or 3D-CAM | assessed up to postoperative day 5 or patient discharge, whichever came first
  Subgroup analysis according to the surgery type, patients' age, and preoperative cognitive function and frailty
Electroencephalography (EEG) | Intraoperative period
  EEG substudy are pre-planned. The association between the development of postoperative delirium, pre&postoperative cognitive function, severe postoperaitve pain and spectral power of alpha, beta, delta, and theta band. Phase-amplitude coupling of each bands

CONTACTS AND LOCATIONS:
Overall Officials: Jiseon jeong, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The dataset generated during the current study is available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Kim J, Lee S, Park B, Sim WS, Ahn HJ, Park MH, Jeong JS. Effect of remimazolam versus propofol anesthesia on postoperative delirium in neurovascular surgery: study protocol for a randomized controlled, non-inferiority trial. Perioper Med (Lond). 2024 Jun 14;13(1):56. doi: 10.1186/s13741-024-00415-6. PMID 38877533